CLINICAL TRIAL: NCT02499081
Title: Phase II Prospective Evaluation of Bone Remodeling During Ixazomib Treatment Relapsed/Refractory Multiple Myeloma Patients
Brief Title: UARK 2014-14: Phase II Prospective Evaluation of Bone Remodeling During Ixazomib Treatment
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Arkansas (Other)
Collaborators: Millennium Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 203444
Record Dates: First submitted 2015-07-09; First posted 2015-07-15 (Estimated); Results first posted 2021-05-14 (Actual); Last update posted 2021-06-11 (Actual); Status verified 2021-04

CONDITIONS: Multiple Myeloma
Keywords: Relapsed; Refractory; Proteasome Inhibitor
MeSH Terms: conditions — Multiple Myeloma; Recurrence | interventions — ixazomib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Ixazomib (Experimental): Ixazomib 4.0 mg given on days 1, 8 15, 22 of a 28 day cycle maximum of 6 cycles.
  Interventions: Drug: Ixazomib

INTERVENTIONS:
Drug: Ixazomib
  Other Names: (MLN 9708)

SUMMARY:
The purpose of this study is to evaluate the effect of Ixazomib on inducing osteoblast activation as measured by bone markers and imaging in patients with relapsed/refractory myeloma.

DETAILED DESCRIPTION:
This is a phase II study designed to examine the bone anabolic effect of the next generation proteasome inhibitor, ixazomib, in relapsed/refractory myeloma patients. Treatment consists of Ixazomib 4 mg on days 1, 8, 15, 22 of a 28 day cycle, for a maximum of 6 cycles. Determination of relapsed/refractory disease as an entry criterion may be based on patient data obtained during or following the patient's most recent prior antineoplastic therapy. Treatment periods will be defined as 28-day cycles. Patients will be seen at regular intervals while they are participating in the study.

ELIGIBILITY:
Inclusion Criteria:

Male or female patients 18 years or older.

* Voluntary written consent must be given before performance of any study related procedure not part of standard medical care, with the understanding that consent may be withdrawn by the patient at any time without prejudice to future medical care.
* Female patients who:

Are postmenopausal for at least 1 year before the screening visit, OR Are surgically sterile, OR If they are of childbearing potential, agree to practice 2 effective methods of contraception, at the same time, from the time of signing the informed consent form through 90 days after the last dose of study drug, AND Agree to practice true abstinence when this is in line with the preferred and usual lifestyle of the subject. (Periodic abstinence [eg, calendar, ovulation, symptothermal, post-ovulation methods] and withdrawal are not acceptable methods of contraception.)

Male patients, even if surgically sterilized (ie, status post-vasectomy), must agree to one of the following:

Agree to practice effective barrier contraception during the entire study treatment period and through 90 days after the last dose of study drug, OR Agree to practice true abstinence when this is in line with the preferred and usual lifestyle of the subject. (Periodic abstinence (eg, calendar, ovulation, symptothermal, post-ovulation methods] and withdrawal are not acceptable methods of contraception.)

* Patients must have a diagnosis of relapsed/refractory multiple myeloma and must have received at least one line of prior therapy.
* Eastern Cooperative Oncology Group (ECOG) performance status and/or other performance status 0, 1, or 2.
* Patients must meet the following clinical laboratory criteria:

Absolute neutrophil count (ANC)1,000/mm3 and platelet count 75,000/mm3. Platelet transfusions to help patients meet eligibility criteria are not allowed within 3 days before study enrollment.

Total bilirubin1.5 the upper limit of the normal range (ULN). Alanine aminotransferase (ALT) and aspartate aminotransferase (AST) 3 ULN. Calculated creatinine clearance 30 mL/min.

Exclusion Criteria:

* Female patients who are lactating or have a positive serum pregnancy test during the screening period.
* Failure to have fully recovered (ie, Grade 1 toxicity) from the reversible effects of prior chemotherapy.
* Major surgery within 14 days before enrollment.
* Radiotherapy within 14 days before enrollment. If the involved field is small (in the opinion of the enrolling investigator), 7 days will be considered a sufficient interval between treatment and administration of the ixazomib.
* Patients who have non-myeloma related bone disease that will interfere with the interpretation of the bone-related blood and radiology assessments, including Paget's disease, Rickets, Osteomalacia, and any other metastatic bone cancer.
* History of myeloma-related central nervous system involvement.
* Infection requiring systemic antibiotic therapy or other serious infection within 14 days before study enrollment.
* Evidence of current uncontrolled cardiovascular conditions, including uncontrolled hypertension, uncontrolled cardiac arrhythmias, symptomatic congestive heart failure, unstable angina, or myocardial infarction within the past 6 months.
* Systemic treatment, within 14 days before the first dose of ixazomib, with strong inhibitors of CYP1A2 (fluvoxamine, enoxacin, ciprofloxacin), strong inhibitors of CYP3A (clarithromycin, telithromycin, itraconazole, voriconazole, ketoconazole, nefazodone, posaconazole) or strong CYP3A inducers (rifampin, rifapentine, rifabutin, carbamazepine, phenytoin, phenobarbital), or use of Ginkgo biloba or St. John's wort.
* Ongoing or active systemic infection, known active hepatitis B or C virus infection, or known human immunodeficiency virus (HIV) positive.
* Any serious medical or psychiatric illness that could, in the investigator's opinion, potentially interfere with the completion of treatment according to this protocol.
* Known allergy to any of the study medications, their analogues, or excipients in the various formulations of any agent.
* Known GI disease or history of GI procedure that could interfere with the oral absorption or tolerance of ixazomib including difficulty swallowing.
* Diagnosed or treated for another malignancy within 2 years before study enrollment or previously diagnosed with another malignancy and have any evidence of residual disease. Patients with non-melanoma skin cancer or carcinoma in situ of any type are not excluded if they have undergone complete resection.
* Patient has Grade 3 peripheral neuropathy, or Grade 2 with pain on clinical examination during the screening period.
* Participation in other clinical trials, including those with other investigational agents not included in this trial, within 21 days of the start of this trial and throughout the duration of this trial.
* Patients who have taken bisphosphonate or RANK Ligand Inhibitor within 3 weeks from screening.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2015-09 (Actual); Primary Completion 2018-05-17 (Actual); Study Completion 2018-05-17 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Maurizio Zangari, MD, Principal Investigator — University of Arkansas
Locations (1):
- University of Arkansas for Medical Science, Little Rock, Arkansas, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Ixazomib
Started | 20
Completed | 1
Not Completed | 19

BASELINE CHARACTERISTICS:
Population: Up to 20 adult patients with confirmed diagnosis of relapsed/refractory multiple myeloma will receive Ixazomib.
Groups:
- Ixazomib: Ixazomib 4.0 mg given on days 1, 8 15, 22 of a 28 day cycle maximum of 6 cycles.
  Ixazomib
Arm/Group | Ixazomib
Number analyzed (Participants) | 20
Age, Continuous [Mean (Standard Deviation); unit: years] | 70.91 (10.27)
Sex/Gender, Customized [Number; unit: participants]
  Male | 11
  Female | 9
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2
  Not Hispanic or Latino | 18
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 2
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 4
  White | 14
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 20

OUTCOME MEASURES:

1. Primary Outcome: Change in Serum Osteocalcin From Baseline to End of Study in Patients With Relapsed/Refractory Multiple Myeloma.
Description: To evaluate the effect of Ixazomib on inducing osteoblast activation as measured by change in serum osteocalcin from baseline to end of study in patients with relapsed/refractory multiple myeloma.
Time Frame: Baseline, Treatment (28-day cycles for 6 cycles)
Measure: Median (95% Confidence Interval); unit: ng/ML
Arm/Group | Ixazomib
Number analyzed (Participants) | 20
ng/ML | 20.00 [17.50 to 25.50]

ADVERSE EVENTS:
Time Frame: Pretreatment Events were collected from Baseline until initiation of study drug. Adverse Events (AEs) were collected from the start of the study drug through the end of study treatment (28-day cycles for 6 cycles or until disease progression/intolerable toxicity).
Description: A Pretreatment Event is any untoward medical occurrence in a patient or subject who has signed informed consent to participate in a study but before administration of any study medication.
  AEs are systematically collected and assessed throughout the study via monitoring clinical symptoms; laboratory, pathological, radiological, or surgical findings; physical exam; or other appropriate tests/procedures. AEs may also be self-reported by the patient.
Arm/Group | Ixazomib
All-Cause Mortality (participants affected / at risk) | 15/20
Serious Adverse Events (participants affected / at risk) | 8/20
Other Adverse Events (participants affected / at risk) | 20/20
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Ixazomib (N=20)
Anemia (Blood and lymphatic system disorders) | 8 (32)
Febrile Neutropenia (Blood and lymphatic system disorders) | 2 (3)
Lymphocyte Count Decreased (Blood and lymphatic system disorders) | 8 (44)
Neutrophil count decreased (Blood and lymphatic system disorders) | 2 (5)
Platelet count decreased (Blood and lymphatic system disorders) | 6 (65)
Wbc decrease (leukopenia) (Blood and lymphatic system disorders) | 2 (16)
Vomiting (Gastrointestinal disorders) | 1 (1)
Pain (Gastrointestinal disorders) | 1 (1)
Hypermagnesemia (Metabolism and nutrition disorders) | 2 (5)
Hypokalemia (Metabolism and nutrition disorders) | 2 (5)
Hyponatremia (Metabolism and nutrition disorders) | 2 (5)
Headache (Nervous system disorders) | 1 (1)
Syncope (Nervous system disorders) | 1 (1)
Anxiety (Psychiatric disorders) | 1 (1)
Hypertension (Vascular disorders) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Ixazomib (N=20)
Anemia (Blood and lymphatic system disorders) | 11 (158)
Lymphocyte count decreased (Blood and lymphatic system disorders) | 5 (64)
Neutrophil count decreased (Blood and lymphatic system disorders) | 4 (11)
Platelet count decreased (Blood and lymphatic system disorders) | 14 (115)
Wbc decrease (leukopenia) (Blood and lymphatic system disorders) | 10 (45)
Ear and labyrinth disorders - Other, specify (Ear and labyrinth disorders) | 1 (1)
Tinnitus (Ear and labyrinth disorders) | 1 (1)
Blurred vision (Eye disorders) | 1 (1)
Dry eye (Eye disorders) | 1 (1)
Eye disorders - other (Eye disorders) | 2 (2)
Photophobia (Eye disorders) | 1 (1)
Watering eyes (Eye disorders) | 2 (2)
Constipation (Gastrointestinal disorders) | 2 (4)
Diarrhea (Gastrointestinal disorders) | 9 (12)
Dyspepsia (Gastrointestinal disorders) | 1 (1)
Gastroesophageal reflux disease (Gastrointestinal disorders) | 1 (1)
Gastrointestinal disorders - Other, specify (Gastrointestinal disorders) | 2 (2)
Nausea (Gastrointestinal disorders) | 9 (9)
Vomiting (Gastrointestinal disorders) | 3 (5)
Chills (General disorders) | 1 (1)
Edema limbs (General disorders) | 1 (1)
Fatigue (General disorders) | 15 (27)
Fever (General disorders) | 1 (1)
Gait disturbance (General disorders) | 1 (1)
Malaise (General disorders) | 1 (1)
Pain (General disorders) | 1 (4)
Alanine aminotransferase increased (Hepatobiliary disorders) | 3 (7)
Alkaline phosphatase increased (Hepatobiliary disorders) | 7 (17)
Aspartate aminotransferase increased (Hepatobiliary disorders) | 4 (14)
Blood bilirubin increased (Hepatobiliary disorders) | 2 (6)
Hypoalbuminemia (Hepatobiliary disorders) | 16 (70)
Infections and infestations - Other, specify (Immune system disorders) | 1 (1)
Upper respiratory infection (Immune system disorders) | 2 (2)
Bruising (Injury, poisoning and procedural complications) | 2 (2)
Anorexia (Metabolism and nutrition disorders) | 1 (1)
Bicarbonate decrease (Metabolism and nutrition disorders) | 7 (15)
Hypercalcemia (Metabolism and nutrition disorders) | 4 (8)
Hyperglycemia (Metabolism and nutrition disorders) | 17 (92)
Hyperkalemia (Metabolism and nutrition disorders) | 1 (2)
Hypocalcemia (Metabolism and nutrition disorders) | 12 (67)
Hypokalemia (Metabolism and nutrition disorders) | 6 (38)
Hypomagnesemia (Metabolism and nutrition disorders) | 1 (1)
Hyponatremia (Metabolism and nutrition disorders) | 8 (54)
Back pain (Musculoskeletal and connective tissue disorders) | 5 (6)
Muscle weakness lower limb (Musculoskeletal and connective tissue disorders) | 1 (1)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 4 (4)
Cognitive disturbance (Nervous system disorders) | 1 (1)
Dizziness (Nervous system disorders) | 6 (6)
Headache (Nervous system disorders) | 3 (4)
Neuralgia (Nervous system disorders) | 1 (1)
Peripheral sensory neuropathy (Nervous system disorders) | 10 (10)
Transient ischemic attacks (Nervous system disorders) | 1 (1)
Tremor (Nervous system disorders) | 1 (1)
Depression (Psychiatric disorders) | 1 (1)
Insomnia (Psychiatric disorders) | 4 (4)
Psychiatric disorders - Other, specify (Psychiatric disorders) | 1 (1)
Creatinine increased (Renal and urinary disorders) | 12 (102)
Renal and urinary disorders - Other, specify (Renal and urinary disorders) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 3 (5)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 4 (5)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Postnasal drip (Respiratory, thoracic and mediastinal disorders) | 5 (6)
Productive cough (Respiratory, thoracic and mediastinal disorders) | 3 (3)
Sleep apnea (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Alopecia (Skin and subcutaneous tissue disorders) | 1 (2)
Dry skin (Skin and subcutaneous tissue disorders) | 1 (1)
Pruritus (Skin and subcutaneous tissue disorders) | 1 (1)
Rash acneiform (Skin and subcutaneous tissue disorders) | 2 (2)
Urticaria (Skin and subcutaneous tissue disorders) | 1 (1)
Hypermagnesemia (Metabolism and nutrition disorders) | 2 (7)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-05-15): https://cdn.clinicaltrials.gov/large-docs/81/NCT02499081/Prot_SAP_001.pdf